CLINICAL TRIAL: NCT07305220
Title: Safety Profile Study of Ultrasound-guided Transparietal Lung Biopsy in Patients With Diffuse Interstitial Lung Disease
Brief Title: Safety Profile of Ultrasound-guided Transparietal Lung Biopsy in Patients With Diffuse Interstitial Lung Disease
Acronym: TOUCANS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DR240161; 2024-A01304-43 (Other: ANSM)
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Lung Disease (ILD)
Keywords: Interstitial Lung Disease (ILD); Transthoracic Ultrasound-Guided Biopsy (BPTE); Safety Assessment; Histological Diagnosis
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Primary Purpose : safety
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transthoracic ultrasound-guided lung biopsy (Experimental): patients with surgical lung biopsy indication validated by MDD
  Interventions: Procedure: Transthoracic ultrasound-guided lung biopsy

INTERVENTIONS:
Procedure: Transthoracic ultrasound-guided lung biopsy — * Scheduled 2-4 weeks before SLB
  * Performed under local anesthesia and spontaneous ventilation
  * Target zone identified via CT and ultrasound (B-lines >3/field or pleural irregularities)
  * Biopsy performed using a specialized needle during brief apnea
  * One or two samples taken depending on quality (>1 cm)

SUMMARY:
Rationale Interstitial lung diseases (ILDs) require accurate histological diagnosis when imaging is inconclusive, yet current techniques-surgical lung biopsy and transbronchial cryobiopsy-carry significant risks and lack real-time guidance. BPTE, widely used in oncology, provides ultrasound-guided sampling under local anesthesia with historically lower complication rates, but its value in ILD remains unproven. The TOUCANS study aims to generate safety and feasibility data to support its potential use as a less invasive diagnostic alternative.

Objectives The primary objective is to assess the safety of BPTE in ILD patients, focusing on major adverse events: death, pneumothorax requiring drainage, hemorrhage requiring intervention, and prolonged pleural drainage. Secondary objectives include evaluating all complications within two months, comparing BPTE histological quality with surgical biopsy, and assessing pain, dyspnea, analgesic use, healing, drainage duration, and hematoma on thoracoscopic imaging.

Materials and Methods Fifteen patients aged 18-75 with ILD requiring tissue diagnosis after multidisciplinary review will be included. Exclusion criteria cover coagulation disorders, severe comorbidities, long-term oxygen therapy, impaired lung function, obesity, pulmonary hypertension, anesthetic allergy, and vulnerable populations. BPTE will be performed 2-4 weeks before surgical biopsy, under local anesthesia and spontaneous ventilation, with CT- and ultrasound-guided targeting. One or two biopsies will be taken, followed by ultrasound and chest X-ray monitoring; discharge occurs after four hours if stable. Surgical thoracoscopic biopsy will then be carried out with standard postoperative care. Pain, dyspnea, healing, and imaging findings will be recorded, and histological samples will be reviewed blindly. Data will be captured in eCRFs according to GDPR/CNIL requirements.

Expected Outcomes TOUCANS will provide the first prospective evidence on BPTE for ILD. Demonstrating safety and adequate diagnostic yield could position BPTE as a minimally invasive, outpatient, ultrasound-guided alternative to surgical biopsy. This may shorten diagnostic pathways, reduce complications, and offer a viable option for patients unsuitable for surgery, ultimately improving early management and prognosis.

DETAILED DESCRIPTION:
The TOUCANS study is a prospective, interventional, single-center protocol designed to evaluate the feasibility and safety of transthoracic ultrasound-guided lung biopsy (BPTE) for the histopathological assessment of patients with interstitial lung disease (ILD). Surgical lung biopsy (SLB) remains the reference diagnostic standard when high-resolution CT and multidisciplinary evaluation are inconclusive; however, SLB requires general anesthesia and thoracoscopy and is associated with non-negligible morbidity. Cryobiopsy offers a less invasive option but still relies on general anesthesia and does not provide real-time guidance during tissue acquisition. BPTE, routinely used in oncology, may provide a safer and more accessible alternative by combining real-time thoracic ultrasound guidance with local anesthesia and outpatient feasibility. Its use in ILD has been limited due to a lack of prospective safety and diagnostic performance data.

Scientific Background ILDs often involve peripheral and subpleural abnormalities that can be visualized using thoracic ultrasound. Real-time ultrasound allows operators to identify pleural irregularities, increased B-lines, or localized reductions in aeration that may correspond to accessible sampling sites. These features form the basis for selecting BPTE target zones. BPTE has shown low complication rates in other clinical contexts, including pneumothorax and hemorrhage, but its applicability to ILD requires systematic evaluation given the underlying fragility of this patient population.

Study Rationale By performing both BPTE and SLB in each participant, the study aims to document the safety profile of BPTE relative to the current gold standard and compare tissue quality. This within-subject design allows direct assessment of histological adequacy and potential concordance between techniques, while limiting inter-individual variability. The protocol also aims to document patient-reported outcomes such as pain and dyspnea and to characterize local tissue effects at the BPTE site during subsequent thoracoscopy.

Study Procedures After standard diagnostic workup and confirmation of biopsy indication by multidisciplinary discussion, participants undergo baseline clinical assessment and high-resolution CT imaging. BPTE is performed 2-4 weeks before SLB to ensure procedural independence and adequate healing time. Under local anesthesia and spontaneous ventilation, the operator identifies an appropriate intercostal window using thoracic ultrasound. A target region is selected based on pleural surface abnormalities or an increased number of B-lines. One or two core biopsies measuring at least 1 cm are obtained using a dedicated cutting needle during a brief apnea. Post-procedure monitoring includes lung ultrasound and chest radiography to detect pneumothorax. Patients are discharged after a four-hour observation period unless complications occur.

SLB is performed under general anesthesia via video-assisted thoracoscopy. The thoracic surgeon documents the BPTE site, enabling evaluation of hematoma or other local effects. Standard postoperative care includes pleural drainage and scheduled follow-up visits. Histological samples obtained through BPTE are stored and analyzed at the end of the follow-up period to ensure blinded comparison with surgical specimens.

Data Collection and Management Clinical assessments include evaluation of procedural tolerance, pain, dyspnea, and healing. Thoracoscopic imaging of the BPTE site provides additional information on local changes. All data are entered into electronic case report forms (eCRFs) with access restricted to authorized study personnel. Data management follows GDPR and CNIL requirements, with predefined monitoring procedures to ensure accuracy, completeness, and consistency.

Statistical Approach Given the exploratory nature of the study, the sample size of 15 participants is based on feasibility considerations. Analyses will primarily rely on descriptive statistics to summarize safety outcomes, histological adequacy, and patient-reported measures. No formal hypothesis testing is planned, but the dataset is expected to support the design of future multicenter studies.

Safety Oversight Adverse events and serious adverse events will be documented throughout the study period. Investigators are responsible for evaluating severity and causality and reporting events to the sponsor. An independent safety monitoring committee will review safety data periodically. Regulatory and ethical compliance includes approval from national authorities and ethics committees, informed consent procedures, and insurance coverage for participants.

Expected Contribution The TOUCANS study will provide the first prospective evidence on BPTE in ILD. The findings may clarify whether BPTE can serve as a safe and technically reliable method for obtaining diagnostic tissue in selected ILD patients, potentially reducing the need for surgical biopsy and improving access to histological diagnosis in those with contraindications to invasive procedures.

ELIGIBILITY:
Inclusion Criteria

* Age 18-75 years
* Diagnosed with diffuse ILD
* Histological analysis required after standard diagnostic workup
* Biopsy indication validated by MDD
* Affiliated with French social security
* Written informed consent Exclusion Criteria
* Contraindication to SLB
* Coagulation disorders
* Significant comorbidities affecting safety
* Long-term oxygen therapy
* FVC <55%, DLCO <40%
* BMI >35 kg/m²
* Pulmonary hypertension (PAPS >40 mmHg)
* Allergy to anesthetics
* Protected populations (pregnant women, minors, legally protected adults)
* β-HCG test required for non-menopausal women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of serious complications between BPTE and SLB | From BPTE to the surgical biopsy (2-4 weeks)
  The study monitors for the following adverse events:
  * Death related to the procedure
  * Pneumothorax requiring pleural drainage
  * Pulmonary or chest wall hemorrhage necessitating medical intervention, such as Blood transfusion, Arterial embolization, Surgical management
  This endpoint is designed to evaluate the safety and feasibility of BPTE as a diagnostic tool, particularly in comparison to more invasive procedures like surgical biopsy. The goal is to determine whether BPTE can be safely performed in an outpatient setting with an acceptable risk profile for serious complications.

SECONDARY OUTCOMES:
All complications up to 2 months | From BPTE to 2-month post-surgical biopsy visit
  Occurrence of any complication, whether serious or not.
Duration of pleural drainage | Between BPTE procedure and surgical biopsy.Between surgical biopsy and 1-month post-surgical biopsy visit.
  Evaluation of the duration of pleural drainage after BPTE (if necessary) and after the surgical biopsy
Histological diagnoses | During BPTE procedure, during surgical biopsy
  Histological diagnoses established from the analysis of the sample obtained by BPTE and from the surgical biopsy sample.
Pain assessment | After BPTE and after surgical biopsy: Evaluation at the end of the procedure, after 1hour, 2hours, 3hours, 4hours, 24hours, 2days, 7days, 14days. At 1-month and 2-month post-surgical biopsy visits.
  Pain will be assessed by Numeric Pain Rating Scale (0 = No pain to 10 = Worst imaginable pain) at the site of the area biopsied by BPTE and at the site of the thoracoscopy scars.
Type of analgesics used | After the BPTE until the surgical biopsy. After the surgical biopsy until the visit at 1 month. At 1-month and 2-month post-surgical biopsy visits.
  Daily collection of the type of analgesic (step 1, 2 or 3) used.
Quantity of analgesics used | From the BPTE until the surgical biopsy. From the surgical biopsy until the one-month visit. During the post-surgery visits at one month and two months.
  Daily collection of the quantity (daily cumulative dose) of analgesics used.
Dyspnea assessment | Just before and after BPTE AND just before and and after surgical biopsy: at the end of the procedure, after 1hour, 2hours, 3hours, 4hours, 24hours, 2days, 7days, 14days. At 1-month and 2-month post-surgical biopsy visits.
  Dyspnea will be assessed by Numeric Dyspnea Rating Scale (0= No shortness of breath to 10 = Worst imaginable shortness of breath)
Hematoma detection | Photograph taken by the surgeon during the surgical biopsy assessed by the pulmonologist during the 2-months post-surgical visit.
  Search for a hematoma in the area of the lung biopsied by BPTE on the photograph taken during the surgical biopsy via thoracoscopiy
Healing assessment at biopsy sites | 1-month and 2-months post-surgical biopsy visits.
  Evaluation of the healing of the BPTE puncture site and the surgical access route - Visible or not
  - If visible, specify the appearance : normal, inflammatory, or infected.

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumology department, Tours, France

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the current study will be made available from the corresponding author on reasonable request. The conditions for the transfer of all or part of the database will be decided by the study sponsor and will be the subject of a written contract.